CLINICAL TRIAL: NCT04723251
Title: The Gratitude Gallery - A Positive Psychology Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Erin Hendriks, Assistant Professor of Family Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00177310
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Depression; Anxiety
Keywords: Photos; Photography; Gratitude
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taking Photographs (Experimental): Participants will be asked to take photos with their cell phone.
  Interventions: Behavioral: taking photographs

INTERVENTIONS:
Behavioral: taking photographs — Participants will photograph images (using a cell phone) that invoke a feeling of gratitude. At least 1 photograph (at any time of the day) should be taken for a period of three weeks.
  Once the photo images are captured, the participant should spend a moment looking at the image and reflecting on why they are grateful for the subject of the photograph.

SUMMARY:
This study will assess the feasibility and acceptability of a positive psychology intervention, The Gratitude Gallery, for increasing gratitude in adults.

The study hypothesizes that participants will find the activity feasible and acceptable and complete the intervention as directed. The project also hypothesizes that those that complete the intervention will show an increase in self-reported gratitude, as well as a decrease in symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Able to read/understand English and give consent
* Owns a smart phone capable of taking pictures
* Willing and able to comply with all aspects of study procedures
* PHQ-9 score greater or equal to 5 but less or equal to 14 with no suicidal ideation
* Generalized anxiety disorder (GAD-7) score greater or equal to 0 but less or equal to 9
* No plan to initiate a new program that could increase positive affect during the study period (e.g., psychotherapy, new exercise regimen, meditation classes)
* If on medication then stable (at least 3 months) on dose or not on medication

Exclusion Criteria:

* Having a psychotic disorder active suicidality or severe depressive or anxiety symptoms
* Other factors that at the discretion of the investigators that would adversely affect study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Acceptability of the The Gratitude Gallery | 2 years
  Number of participants that are eligible for the study compared to the number of patients that are enrolled. The higher the ratio of participants enrolled the higher acceptability.
Feasibility of the The Gratitude Gallery | up to 21 days (days of treatment)
  Participants that complete 15 of the 21 intervention days will be considered to be feasible.
Changes in the level of reported gratitude as measured by the Gratitude Questionnaire - 6 (GQ-6). | Baseline, up to day 60
  This is a six question, self-reported survey designed to assess individual differences in the proneness to experience gratitude in daily life. The GQ-6 uses a 7-point Likert scale with responses that range from "strongly disagree" to "strongly agree". Questions 3 and 6 are reverse scored. A higher total score indicated higher levels of gratitude.

SECONDARY OUTCOMES:
Changes in positive and negative affect as measured by the Positive and Negative Affect Scale (PANAS) Scale | Baseline, up to day 60
  The PANAS scale is a 20 item mood scale measuring the two primary dimensions of mood. Responses on a 5-point Likert Scale range from "very slightly or not at all" to "extremely". Positive affect and negative affect questions are grouped and scored separately. The PANAS has been shown to be sensitive to short-term fluctuations in mood in addition to showing stability over a longer (2-month) time period.
Changes in General Life Satisfaction - Fixed Form B from the NIH Toolbox | Baseline, up to day 60
  This is a brief 5-item questionnaire which can be administered to adults over the age of 18. It uses a 7-point Likert scale with responses that range from "strongly disagree" to "strongly agree". The scores for each question are added to create a raw score. This raw score is then converted to a T-score using a conversion table which represents the mean of the United States population.
Changes in sleep quality using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance - Short Form 4a | Baseline, up to day 60
  This assessment consists of 4 items which measure sleep quality and sleep disturbances using a 5 point likert scale ranging in value from 1 to 5 with higher scores indicating greater sleep quality.
Changes in depressive symptoms using the Patient Health Questionnaire 9-Item (PHQ-9) | Baseline, up to day 60
  The PHQ-9 is a brief, self-administered questionnaire that scores each of the Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria for depression on a scale from 0 to 3. Response options include "not at all", "several days", more than half the days" and "nearly every day". It is a validated measure of depression severity. Scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe, and severe depression, respectively.
Changes in anxiety symptoms using the Generalized Anxiety scale (GAD-7) | Baseline, up to day 60
  The GAD-7 is a self-reported questionnaire that assesses for the seven core symptoms of generalized anxiety disorder and severity. Response options include "not at all", "several days", more than half the days" and "nearly every day". GAD-7 total score for the seven items ranges from 0 to 21. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hendriks, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No